CLINICAL TRIAL: NCT07206212
Title: Efficacy and Cost-effectiveness of a Lifestyle Intervention to Reduce Cardiometabolic Risk Factors in Individuals With Obsessive-compulsive Disorder: A Randomized Controlled Trial
Brief Title: A Lifestyle Intervention to Reduce Cardiometabolic Risk Factors in Individuals With Obsessive-compulsive Disorder
Acronym: LIFT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Lorena Fernández de la Cruz, PhD, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2025-04734-01; 20210493, 20220899 (Other Grant/Funding Number: Swedish Heart and Lung Foundation); 2022-005109 (Other Grant/Funding Number: Swedish Research Council); 2019-00438 (Other Grant/Funding Number: Swedish ResearchCouncil for Health, Working Life and Welfare); 20200139 (Other Grant/Funding Number: Region Stockholm); 2020-01361, 2022-01675 (Other Grant/Funding Number: Karolinska Institutet)
Record Dates: First submitted 2025-09-11; First posted 2025-10-03 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Obsessive Compulsive Disorder (OCD); Lifestyle (Sedentary Behavior and Physical Activity)
Keywords: OCD; Obsessive-compulsive disorder; Cardiovascular disease; Metabolic syndrome; Prevention; Lifestyle habits; Physical activity
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Sedentary Behavior; Motor Activity; Cardiovascular Diseases; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active intervention (Experimental): The lifestyle intervention (LIFT) consists of one initial individual session to create a personal plan and set up goals for a change of lifestyle habits (week 1) and 12 weekly group sessions (weeks 2 to 13) including both education on lifestyle habits and physical exercise. After week 13, participants get access to a booster module in a digital platform to help them maintain their behavioral changes.
  Interventions: Behavioral: A group-based lifestyle intervention for individuals with OCD
- Medical and lifestyle advice (Active Comparator): Participants in this arm will receive one individual session where participants will receive feedback based on the baseline evaluation of their clinical characteristics, lifestyle habits, and cardiometabolic risk (week 1). Additionally, participants will receive written educational information on healthy lifestyle habits.
  Interventions: Behavioral: Medical and lifestyle advice

INTERVENTIONS:
Behavioral: A group-based lifestyle intervention for individuals with OCD — Participants will take part in 13 week program, with one individual session to set up goals for a change of lifestyle habits, based on the baseline evaluation of their clinical characteristics, lifestyle habits, and cardiometabolic risk, and 12 group sessions, consisting of both education on lifestyle habits and physical exercise.
  Each educational session will focus on a specific topic/lifestyle habit, alternating more informative sessions with sessions discussing how the information can be applied, taking into account specific hinders due to Obsessive-Compulsive Disorder.
  Between-sessions homework will include, for example, daily registration of physical activity and implementing changes in the lifestyle habits discussed during each session. All homework assignments will be registered in a digital platform. After the 13 weeks of lifestyle intervention, participants will get access to a booster module in the digital platform to help them maintain their behavioral changes.
  Other Names: LIFT
  Arms: Active intervention
Behavioral: Medical and lifestyle advice — One individual session with a clinical psychologist on week 1 of about 1 hour of duration. During this session, participants will receive feedback based on the baseline evaluation of their clinical characteristics, lifestyle habits, and cardiometabolic risk. Participants also receive written educational information on healthy lifestyle habits based on national Swedish guidelines issued by the National Board of Health and Welfare. The recommendations include engaging in regular physical activity, dietary guidelines based on Nordic Nutrition Recommendations, and advice to reduce alcohol consumption and quit tobacco use.
  Arms: Medical and lifestyle advice

SUMMARY:
The overall aim of this study is to evaluate the efficacy and cost-effectiveness of a lifestyle intervention to improve lifestyle habits and reduce cardiometabolic risk factors in individuals with obsessive-compulsive disorder (OCD).

DETAILED DESCRIPTION:
Obsessive-compulsive disorder (OCD) is a prevalent and impairing disorder with an increased risk of morbidity and mortality due to cardiometabolic diseases. These risks remain significant over and above psychiatric comorbidities and shared familial factors, indicating that at least part of this risk could be a consequence of pernicious lifestyle habits (e.g., physical inactivity, unhealthy diet). A lifestyle intervention targeting cardiometabolic risk factors in people with OCD has previously been deemed feasible, acceptable, and safe. However, the efficacy and cost-effectiveness of the intervention need to be investigated. This will be the first RCT to examine the effects of a lifestyle intervention on the health and well-being of people with OCD.

The specific aims are:

1. to investigate whether the intervention, compared to medical and lifestyle advice (control), is effective in increasing physical activity (objectively measured with an accelerometer);
2. to investigate the efficacy of the intervention, vs. the control, in changing cardiometabolic risk factors (lifestyle habits, cardiometabolic physiological, and laboratory measurements), mental health measures, functional impairment, and quality of life; and
3. to evaluate whether the lifestyle intervention, vs. the control, is cost-effective from a healthcare provider perspective.

ELIGIBILITY:
Inclusion criteria:

1. A diagnosis of obsessive-compulsive disorder (OCD), based on the diagnostic criteria of the 5th edition of the Diagnostic and Statistical Manual of Mental Disorders. Screened at registration and at the initial phone call and confirmed by the assessor at the inclusion assessment (psychiatric interview), using a semi-structured diagnostic interview.
2. Physical inactivity/sedentarism, operationalized as less than 150 minutes of physical activity per week during the last month, evaluated by asking two questions from the Swedish National Board of Health and Welfare concerning 1) frequency of weekly moderate or vigorous intensity physical exercise and 2) frequency of weekly non-exercise/daily life physical activity. Screened at registration and at the initial phone call and confirmed by the assessor at the inclusion assessment (psychiatric interview).
3. Aged 18 years or older. Screened at registration and confirmed by the assessor at the initial phone call and/or confirmed by the assessor at the inclusion assessment (psychiatric interview).

Exclusion criteria:

1. Intellectual disability or severe psychiatric symptoms or suicidal risk that could interfere with the intervention. Screened at the initial phone call and confirmed by the assessor at the inclusion assessment (psychiatric interview), using a semi-structured diagnostic interview.
2. A diagnosis of an eating disorder or a substance use disorder. Screened at the initial phone call and confirmed by the assessor at the inclusion assessment (psychiatric interview), using a semi-structured diagnostic interview.
3. Being pregnant or <1 year postpartum. Screened at the initial phone call and confirmed by the assessor at the inclusion assessment (psychiatric interview).
4. Myocardial infarction or stroke within the last 6 months. Screened at registration and confirmed by the assessor at the initial phone call and/or the inclusion assessment (physiological measures).
5. Cardiovascular risk measures significantly over the normal range (e.g., severe hypertension [blood pressure above ≥180 mmHg systolic or ≥110 mmHg diastolic]) or a current somatic condition that make participation in the intervention contraindicated. Screened at registration and confirmed by the assessor at the initial phone call and/or the inclusion assessment (physiological measures), after consulting with the study doctor, if necessary.
6. Initiation or adjustment of any cardiometabolic medication (e.g., blood pressure or blood lipids lowering mediation) within 3 months prior to assessments. Screened at registration and confirmed by the assessor at the initial phone call and/or the inclusion assessment (physiological measures).
7. Inability to understand and communicate in Swedish. Confirmed by the assessor at the initial phone call.
8. Inability to consistently attend the sessions involved in the intervention. Screened by the assessor at the initial phone call and/or confirmed by the assessor at the inclusion assessment (psychiatric interview).
9. Inability to travel to the sessions involved in the intervention. Screened by the assessor at the initial phone call and/or confirmed by the assessor at the inclusion assessment (psychiatric interview).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2026-01-30 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Physical activity: Steps per day | Baseline, week 14 after the start of the intervention (primary endpoint), 3 months after the primary endpoint, 6 months after the primary endpoint, 12 months after the primary endpoint.
  Measured as change in steps/day with an accelerometer. Participants will be asked to wear an accelerometer (activPAL™) 24 hours/day for seven consecutive days at each assessment point. The device is placed on the thigh. Data will be considered valid if wear time is ≥10 hours/day for at least 4 days, including at least one weekend day.

SECONDARY OUTCOMES:
Physical activity: Moderate to vigorous physical activity (MVPA) | Baseline, week 14 after the start of the intervention (primary endpoint), 3 months after the primary endpoint, 6 months after the primary endpoint, 12 months after the primary endpoint.
  MVPA per day operationalised as a walking cadence of >100 steps/minute.
International Physical Activity Questionnaire, short form (IPAQ-SF) | Baseline, week 14 after the start of the intervention (primary endpoint), 3 months after the primary endpoint, 6 months after the primary endpoint, 12 months after the primary endpoint.
  Self-reported assessment of physical activity (moderately intense activities, vigorously intense activities, walking) and sedentary time during the last 7 days. Responses on each physical activity intensity question will be converted to metabolic equivalent of task (MET) minutes, using the formula from the IPAQ scoring protocol. Both the continuous and categorical scores (high, moderate, and low) will be calculated according to the scoring guidelines. A higher MET score corresponds to higher levels of physical activity.
15-item Food Frequency Questionnaire (FFQ) | Baseline, week 14 after the start of the intervention (primary endpoint), 3 months after the primary endpoint, 6 months after the primary endpoint, 12 months after the primary endpoint.
  Self-reported assessment of dietary patterns. It consists of 15 items concerning dietary choices, where each item is evaluated as either meeting or not meeting the guidelines set in the Nordic Nutrition Recommendations (NNR). Each met recommendation receives 1 point, resulting in a healthy eating index ranging from 0 to 15 points. Based on this index, dietary patterns are classified as good (9 or more points), average (6-8 points) or poor (5 or fewer points).
Alcohol Use Disorder Identification Test for Consumption (AUDIT-C) | Baseline, week 14 after the start of the intervention (primary endpoint), 3 months after the primary endpoint, 6 months after the primary endpoint, 12 months after the primary endpoint.
  Self-reported assessment of alcohol consumption. Scores in the AUDIT-C range from 0 to 12 points, where 0 points indicate no alcohol use. Cut-off scores for risk consumption vary across settings and population, but a score ≥4 points has been suggested as a cut-off for detecting risk consumption of alcohol when validated in the general population.
Tobacco use | Baseline, week 14 after the start of the intervention (primary endpoint), 3 months after the primary endpoint, 6 months after the primary endpoint, 12 months after the primary endpoint.
  Evaluated by asking self-reported questions about current or previous use of cigarettes, snus or other tobacco or nicotine products. If current use, or if they quit during the last 6 months, participants are asked to specify frequency (daily, sometimes) and amount used.
Perceived Stress Scale (PSS) | Baseline, week 14 after the start of the intervention (primary endpoint), 3 months after the primary endpoint, 6 months after the primary endpoint, 12 months after the primary endpoint.
  Self-reported assessment of perceived stress. The total score ranges from 0 to 40, with higher scores indicating higher levels of perceived stress.
Insomnia Severity Scale (ISI) | Baseline, week 14 after the start of the intervention (primary endpoint), 3 months after the primary endpoint, 6 months after the primary endpoint, 12 months after the primary endpoint.
  Self-reported assessment of sleep problems and severity of symptoms. Consists of 7 items that are rated on a 5-point Likert scale to evaluate sleep problems and severity of symptoms. The total score ranges from 0 to 28 points, with a higher score indicating more severe sleep problems.
Yale-Brown Obsessive Compulsive Scale (Y-BOCS) | Baseline, week 14 after the start of the intervention (primary endpoint), 3 months after the primary endpoint, 6 months after the primary endpoint, 12 months after the primary endpoint.
  Clinician-rated semi-structured interview to assess OCD symptom severity. The Y-BOCS consists of 10 items rated from 0 to 4, with a total score from 0 to 40, where a higher score corresponds to more severe OCD.
Obsessive-Compulsive Inventory - 12 (OCI-12) | Baseline, week 14 after the start of the intervention (primary endpoint), 3 months after the primary endpoint, 6 months after the primary endpoint, 12 months after the primary endpoint.
  Self-reported assessment of OCD symptoms. Consists of 12 items rated on a 5-point Likert scale, with total scores ranging from 0-48. Scores between 0 and 12 indicate mild, between 13 and 21 indicate moderate, and between 22 and 48 indicate severe OCD symptoms.
Patient Health Questionnaire (PHQ-9) | Baseline, week 14 after the start of the intervention (primary endpoint), 3 months after the primary endpoint, 6 months after the primary endpoint, 12 months after the primary endpoint.
  Self-reported assessment of symptoms of depression. In this 9-item scale the total score ranges from 0 to 27 points, with a higher score corresponding to more severe symptoms of depression.
EuroQol five dimensional five level questionnaire (EQ-5D-5L) | Baseline, week 14 after the start of the intervention (primary endpoint), 3 months after the primary endpoint, 6 months after the primary endpoint, 12 months after the primary endpoint.
  Self-rated assessment of own health status in five dimensions (mobility; self-care; usual activities; pain/discomfort; and anxiety/depression), within five levels of severity (no problems; slight problems; moderate problems; severe problems; or extreme problems). The scale also comprises a rating of their overall health status on a scale from 0-100 (0 = worst imaginable health; 100 = best imaginable health), the EQ-VAS scale. The scores are combined to calculate a health utility number, with the health utilities ranging from -0.31 for the worst to 1 for the best EQ-5D-5L states in Sweden.
Work and Social Adjustment Scale (WSAS) | Baseline, week 14 after the start of the intervention (primary endpoint), 3 months after the primary endpoint, 6 months after the primary endpoint, 12 months after the primary endpoint.
  Self-reported assessment of impairment in functioning, in terms of work, home management, social leisure activities, private leisure activities, and relationships. Each item is rated on a scale from 0 to 8, with the total score ranging from 0 to 40. A higher score corresponds to more impairment in functioning.
Waist circumference | Baseline, week 14 after the start of the intervention (primary endpoint), 3 months after the primary endpoint, 6 months after the primary endpoint, 12 months after the primary endpoint.
  Measured in a standing position, midway between the lower rib margin and the iliac crest, in centimeters (cm) at the nearest 0.5 cm.
Sagittal abdominal diameter | Baseline, week 14 after the start of the intervention (primary endpoint), 3 months after the primary endpoint, 6 months after the primary endpoint, 12 months after the primary endpoint.
  Measured in a supine position at the nearest 0.1 centimeter with a ruler and a water lever or a caliper, at the level of the umbilical.
Weight | Baseline, week 14 after the start of the intervention (primary endpoint), 3 months after the primary endpoint, 6 months after the primary endpoint, 12 months after the primary endpoint.
  Measured in kilograms, to the nearest 0.1 kg.
Body Mass Index (BMI) | Baseline, week 14 after the start of the intervention (primary endpoint), 3 months after the primary endpoint, 6 months after the primary endpoint, 12 months after the primary endpoint.
  Derived by dividing weight (in kilograms measured to the nearest 0.1 kg) by height (in meters measured to the nearest 0.1 cm) squared.
Systolic and diastolic blood pressure | Baseline, week 14 after the start of the intervention (primary endpoint), 3 months after the primary endpoint, 6 months after the primary endpoint, 12 months after the primary endpoint.
  Measured in a seated position after ten minutes of rest, with a standard sphygmomanometer. The measurement will be taken twice with 1 minute between measures, according to the gold standard for measuring blood pressure.
Resting heart rate | Baseline, week 14 after the start of the intervention (primary endpoint), 3 months after the primary endpoint, 6 months after the primary endpoint, 12 months after the primary endpoint.
  Measured in a seated position following a 5 minute rest.
Total cholesterol | Baseline, week 14 after the start of the intervention (primary endpoint), 3 months after the primary endpoint, 6 months after the primary endpoint, 12 months after the primary endpoint.
  Blood will be drawn following an overnight fast (minimum 8 hours, or else rescheduled). Measured as mmol/l.
S-low density lipoprotein cholesterol | Baseline, week 14 after the start of the intervention (primary endpoint), 3 months after the primary endpoint, 6 months after the primary endpoint, 12 months after the primary endpoint.
  Blood will be drawn following an overnight fast (minimum 8 hours, or else rescheduled). Measured as mmol/l.
S-high density lipoprotein cholesterol | Baseline, week 14 after the start of the intervention (primary endpoint), 3 months after the primary endpoint, 6 months after the primary endpoint, 12 months after the primary endpoint.
  Blood will be drawn following an overnight fast (minimum 8 hours, or else rescheduled). Measured as mmol/l.
Lipoprotein (a) | Baseline, week 14 after the start of the intervention (primary endpoint), 3 months after the primary endpoint, 6 months after the primary endpoint, 12 months after the primary endpoint.
  Blood will be drawn following an overnight fast (minimum 8 hours, or else rescheduled). Measured as nmol/l.
Fasting triglycerides | Baseline, week 14 after the start of the intervention (primary endpoint), 3 months after the primary endpoint, 6 months after the primary endpoint, 12 months after the primary endpoint.
  Blood will be drawn following an overnight fast (minimum 8 hours). Measured as mmol/l.
Fasting plasma glucose | Baseline, week 14 after the start of the intervention (primary endpoint), 3 months after the primary endpoint, 6 months after the primary endpoint, 12 months after the primary endpoint.
  Blood will be drawn following an overnight fast (minimum 8 hours). Measured as mmol/l.
Glycated hemoglobin | Baseline, week 14 after the start of the intervention (primary endpoint), 3 months after the primary endpoint, 6 months after the primary endpoint, 12 months after the primary endpoint.
  Blood will be drawn following an overnight fast (minimum 8 hours) (HbA1c, mmol/l). It reflects average plasma glucose over the previous 8-12 weeks.
Thyroid stimulating hormone (TSH) | Baseline, week 14 after the start of the intervention (primary endpoint), 3 months after the primary endpoint, 6 months after the primary endpoint, 12 months after the primary endpoint.
  Blood will be drawn following an overnight fast (minimum 8 hours). Measured as mE/L.
Cobalamin | Baseline, week 14 after the start of the intervention (primary endpoint), 3 months after the primary endpoint, 6 months after the primary endpoint, 12 months after the primary endpoint.
  Blood will be drawn following an overnight fast (minimum 8 hours). Reflects vitamin B12 status. Measured in pmol/L.
Homocysteine | Baseline, week 14 after the start of the intervention (primary endpoint), 3 months after the primary endpoint, 6 months after the primary endpoint, 12 months after the primary endpoint.
  Blood will be drawn following an overnight fast (minimum 8 hours). Measured in µmol/L.
25-OHD-vitamin | Baseline, week 14 after the start of the intervention (primary endpoint), 3 months after the primary endpoint, 6 months after the primary endpoint, 12 months after the primary endpoint.
  Blood will be drawn following an overnight fast (minimum 8 hours). Main marker of vitamin D status in the body, reported in nmol/L.
Folate | Baseline, week 14 after the start of the intervention (primary endpoint), 3 months after the primary endpoint, 6 months after the primary endpoint, 12 months after the primary endpoint.
  Blood will be drawn following an overnight fast (minimum 8 hours). Reported in nmol/L.
Iron deposits: Iron | Baseline, week 14 after the start of the intervention (primary endpoint), 3 months after the primary endpoint, 6 months after the primary endpoint, 12 months after the primary endpoint.
  Blood will be drawn following an overnight fast (minimum 8 hours). Iron [Fe], reported in µmol/L.
Iron deposits: Transferrin | Baseline, week 14 after the start of the intervention (primary endpoint), 3 months after the primary endpoint, 6 months after the primary endpoint, 12 months after the primary endpoint.
  Blood will be drawn following an overnight fast (minimum 8 hours). Reported in µg/L.
High-sensitive C-reactive protein (CRP) | Baseline, week 14 after the start of the intervention (primary endpoint), 3 months after the primary endpoint, 6 months after the primary endpoint, 12 months after the primary endpoint.
  Blood will be drawn following an overnight fast (minimum 8 hours). Reported in mg/L.
White blood cell telomere length | Baseline, week 14 after the start of the intervention (primary endpoint).
  Blood will be drawn following an overnight fast (minimum 8 hours). Telomere length in leukocytes will be measured, reported as relative telomere length (T/S ratio).
Inflammation panel | Baseline, week 14 after the start of the intervention (primary endpoint).
  Blood will be drawn following an overnight fast (minimum 8 hours). Immune activity plasma proteins (n=92) will be analysed using the Olink Target 96 Inflammation panel.
Extracellular vesicles (EVs) | Baseline, week 14 after the start of the intervention (primary endpoint).
  Blood will be drawn following an overnight fast (minimum 8 hours). EVs will be isolated from plasma using differential ultracentrifugation. Quantification and separation of EVs will be performed using flow cytometry using antibodies specifically marking EVs with regards to being a microparticle and their tissue of origin. We will investigate the amount and origin of EVs from the vascular endothelium, leukocytes, platelets, and the skeletal muscle. To assess the cargo of particularly interesting EVs, RNA will be isolated and miRNA profiled using the robust and high-throughput nCounter (Nanostring).
Biological age | Baseline, week 14 after the start of the intervention (primary endpoint).
  Blood will be drawn following an overnight fast (minimum 8 hours). DNA will be extracted using the Chemagen kits on the Hamilton ChemagicSTAR® platform. Bisulfite conversion will be conducted using the EZ-96 DNA Methylation-Lightning Kit (D5033). The Illumina Infinium MethylationEPIC v.2 array will be used to quantify DNAm at ~930,000 sites. Raw methylation data will be pre-processed using standard quality control steps, including removal of low-quality probes (e.g., detection p-value >0.01), background correction, and normalization. Biological aging patterns will be assessed through epigenetic age calculations using state-of-the-art algorithms (e.g., GrimAge). Accelerated biological age will be calculated as the residual from regressing epigenetic age on chronological age.

OTHER OUTCOMES:
Adverse events | Week 7 after the start of the intervention, week 14 after the start of the intervention (primary endpoint).
  Measured with a short questionnaire created by the research team regarding potential adverse events (e.g., increased anxiety, headaches, increased tiredness, musculoskeletal pain). They will also be able to write own examples on negative experiences connected to participation in the intervention.
Concurrent interventions | Baseline, week 7 after the start of the intervention, week 14 after the start of the intervention (primary endpoint), 3 months after the primary endpoint, 6 months after the primary endpoint, 12 months after the primary endpoint.
  At each measurement point, information will be collected on any treatment changes (e.g., changes in medication, initiation of psychological treatment) and/or initiation of concurrent interventions to improve lifestyle habits (including e.g., vitamin supplements) or cardiometabolic risk factors.

CONTACTS AND LOCATIONS:
Overall Officials: Lorena Fernández de la Cruz, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- OCD-Programmet, Psykiatri Sydväst, Huddinge, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No
The investigators may potentially share trial data from the study with other researchers around the world. The use would primarily be to combine outcome data for potential meta-analyses in this research field. Shared data will be pseudonymised. The possibility of future data sharing is mentioned in the informed consent form.